CLINICAL TRIAL: NCT02485483
Title: Validation of Standardized Questionnaires on Depression for Rheumatoid Arthritis (RA) (VADERA I) and Investigation of the Frequency of Depression in RA (VADERA II)
Brief Title: Study for Validation of Standardized Questionnaires on Depression and Investigation of the Frequency of Depression in Rheumatoid Arthritis (RA) Participants
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Chugai Pharmaceutical (Industry)
Responsible Party: Sponsor
Other Study IDs: ML29326
Record Dates: First submitted 2015-06-26; First posted 2015-06-30 (Estimated); Results first posted 2016-10-17 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-08

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Time Perspective: Prospective

GROUPS / COHORTS (2):
- VADERA I: RA participants without a concurrent history of depression and who have not received psychotherapy, antidepressants, or inpatient psychiatric treatment in the 3 months before baseline (T0) will be asked to complete the World Health Organization Five Well-Being Index (WHO-5), Patient Health Questionnaire-9 (PHQ-9) and Beck Depression Inventory (2nd edition) (BDI-II) questionnaires and a subsequent structured interview using Montgomery-Åsberg Depression Rating Scale (MADRS) at 2 time-points (T0 and T1 [12 ± 2 weeks]) with a 10-14 week interval between assessments.
- VADERA II: All RA participants who are able to complete the PHQ-9 and BDI-II questionnaires, and have been scheduled for a RA consultation at one of the participating clinics will be eligible for participation.

SUMMARY:
The purpose of this study is to validate standardized questionnaires on depression for RA and to investigate the frequency of depression with RA. The study will include 2 parts, VADERA I and VADERA II. In VADERA I, 300 participants will be surveyed twice at an interval of 3 months regarding their current emotional condition using standardized questionnaires. On the basis of the results of VADERA I, in VADERA II, the selected questionnaire will be used to assess the prevalence of depression with RA in approximately 1000 participants.

DETAILED DESCRIPTION:
VADERA I is regarded as interventional epidemiologic study. The study was considered as interventional because of the use of the questionnaires and interview for the diagnosis of depression. VADERA II is a cross-sectional epidemiologic study.

ELIGIBILITY:
Inclusion Criteria:

* VADERA I: Participants diagnosed with RA, who did not suffer from a concurrent, manifest depressive disorder and had been scheduled for a RA consultation at one of the participating clinics
* VADERA II: All participants diagnosed with RA who were able to complete the questionnaires and had been scheduled for a RA consultation at one of the participating clinics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: VADERA I was conducted in 9 clinical centers across Germany. VADERA II was conducted in 10 centers representing the spectrum of clinical settings in Germany where participants are diagnosed with rheumatoid arthritis and included large academic medical centers, community hospitals and private rheumatology practices across Germany.
Sampling Method: Non-Probability Sample
Enrollment: 1292 (Actual)
Dates: Start 2012-11; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (9):
- Germany (9):
  - Berlin
  - Dresden
  - Erlangen
  - Frankfurt
  - Leipzig
  - München
  - Osnabrück
  - Rostock
  - Würzburg

REFERENCES:
- [Derived] Englbrecht M, Alten R, Aringer M, Baerwald CG, Burkhardt H, Eby N, Flacke JP, Fliedner G, Henkemeier U, Hofmann MW, Kleinert S, Kneitz C, Kruger K, Pohl C, Schett G, Schmalzing M, Tausche AK, Tony HP, Wendler J. New insights into the prevalence of depressive symptoms and depression in rheumatoid arthritis - Implications from the prospective multicenter VADERA II study. PLoS One. 2019 May 28;14(5):e0217412. doi: 10.1371/journal.pone.0217412. eCollection 2019. PMID 31136632
- [Derived] Englbrecht M, Alten R, Aringer M, Baerwald CG, Burkhardt H, Eby N, Fliedner G, Gauger B, Henkemeier U, Hofmann MW, Kleinert S, Kneitz C, Krueger K, Pohl C, Roske AE, Schett G, Schmalzing M, Tausche AK, Peter Tony H, Wendler J. Validation of Standardized Questionnaires Evaluating Symptoms of Depression in Rheumatoid Arthritis Patients: Approaches to Screening for a Frequent Yet Underrated Challenge. Arthritis Care Res (Hoboken). 2017 Jan;69(1):58-66. doi: 10.1002/acr.23002. PMID 27482854

RESULTS

PARTICIPANT FLOW:
Groups:
- VADERA I: Rheumatoid arthritis (RA) participants without a concurrent history of depression and who had not received psychotherapy, antidepressants, or inpatient psychiatric treatment in the 3 months before baseline (T0) were asked to complete the World Health Organization Five Well-Being Index (WHO-5), Patient Health Questionnaire-9 (PHQ-9) and Beck Depression Inventory (2nd edition) (BDI-II) questionnaires and a subsequent structured interview using Montgomery-Åsberg Depression Rating Scale (MADRS) at 2 time-points (T0 and T1 [12 ± 2 weeks]) with a 10-14 week interval between assessments.
- VADERA II: All RA participants who were able to complete the PHQ-9 and BDI-II questionnaires, and had been scheduled for a RA consultation at one of the participating clinics were eligible for participation.
Period: Overall Study
Arm/Group | VADERA I | VADERA II
Started | 277 | 1015
Completed | 223 | 1015
Not Completed | 54 | 0
Not completed — Depression at baseline | 15 | 0
Not completed — Discontinued after baseline | 39 | 0

BASELINE CHARACTERISTICS:
Population: All VADERA I and VADERA II participants who had given informed consent and entered into the study database.
Groups:
- VADERA I: RA participants without a concurrent history of depression and who had not received psychotherapy, antidepressants, or inpatient psychiatric treatment in the 3 months before baseline (T0) were asked to complete the WHO-5, PHQ-9 and BDI-II questionnaires and a subsequent structured interview using MADRS at 2 time-points (T0 and T1 [12 ± 2 weeks]) with a 10-14 week interval between assessments.
- Total: Total of all reporting groups
Arm/Group | VADERA I | VADERA II | Total
Number analyzed (Participants) | 277 | 1015 | 1292
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (13.0) | 61.0 (12.9) | 60.7 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 218 | 764 | 982
  Male | 59 | 251 | 310

OUTCOME MEASURES:

1. Primary Outcome: PHQ-9 Score at Baseline: VADERA I
Description: The PHQ-9 is a self-reported questionnaire measuring depressive symptoms.This is a nine item measure with a response score for each item on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). Thus, the total score ranges from 0 to 27; with 0-4 being minimum indicating no depressive symptoms, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-27 severe depression.
Time Frame: Baseline
Population: Validation analysis set of VADERA I population defined as all study participants diagnosed with RA, who had given informed consent, and had no documented depression at baseline. Number of participants analyzed = participants with PHQ-9 score assessment at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | VADERA I
Number analyzed (Participants) | 223
scores on a scale | 5.2 (4.0)
Statistical Analysis 1: Comparison: VADERA I; Number of participants analyzed (N) = 221; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Convergent Validity Criterion Correlation coefficient (ρ) > |0.50|; Spearman correlation coefficient = 0.67, 95% CI 2-sided [0.59 to 0.74] — Convergent correlation between PHQ-9 and MADRS
Statistical Analysis 2: Comparison: VADERA I; Number of participants analyzed (N) = 222; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Convergent Validity Criterion ρ > |0.50|; Spearman correlation coefficient = 0.69, 95% CI 2-sided [0.62 to 0.76] — Convergent correlation between PHQ-9 and BDI-II

2. Primary Outcome: PHQ-9 Score at Week 12 ± 2: VADERA I
Description: The PHQ-9 is a self-reported questionnaire measuring depressive symptoms. This is a nine item measure with a response score for each item on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). Thus, the total score ranges from 0 to 27; with 0-4 being minimum indicating no depressive symptoms, 5-9 mild depression, 10-14 moderate depression, 15-19 moderately severe depression, 20-27 severe depression.
Time Frame: Week 12 ± 2
Population: Validation analysis set of VADERA I population. Number of participants analyzed = participants with PHQ-9 score assessment at specified time-point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | VADERA I
Number analyzed (Participants) | 207
scores on a scale | 4.8 (4.2)
Statistical Analysis 1: Comparison: VADERA I; Number of participants analyzed (N) = 203; Test type: Superiority or Other; p = 0.057, t-test, 2 sided — Convergent Validity Criterion ρ > |0.50|; Spearman correlation coefficient = 0.58, 95% CI 2-sided [0.48 to 0.66] — Convergent correlation between PHQ-9 and MADRS
Statistical Analysis 2: Comparison: VADERA I; Number of participants analyzed (N) = 200; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Convergent Validity Criterion ρ > |0.50|; Spearman correlation coefficient = 0.74, 95% CI 2-sided [0.67 to 0.80] — Convergent correlation between PHQ-9 and BDI-II

3. Primary Outcome: BDI-II Score at Baseline: VADERA I
Description: BDI-II Scale is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represents a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe). Scores for each symptom are added up to obtain the total scores for all 21 items. Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 is minimal depression, 14-19 is mild depression, 20-28 is moderate depression and 29-63 is severe depression.
Time Frame: Baseline
Population: Validation analysis set of VADERA I population. Number of participants analyzed = participants with BDI-II score assessment at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | VADERA I
Number analyzed (Participants) | 261
scores on a scale | 9.3 (7.6)
Statistical Analysis 1: Comparison: VADERA I; Number of participants analyzed (N) = 258; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Convergent Validity Criterion ρ > |0.50|; Spearman correlation coefficient = 0.73, 95% CI 2-sided [0.67 to 0.79] — Convergent correlation between BDI-II and MADRS

4. Primary Outcome: BDI-II Score at Week 12 ± 2: VADERA I
Description: BDI-II Scale is a 21-item self-reported questionnaire which measures the existence and severity of symptoms of depression. Each of the 21 items on BDI-II tool represent a depressive symptom. The symptoms are each scored on a 4-point Likert scale of 0 to 3 (0=symptom is absent; 3=symptom is severe). Scores for each symptom are added up to obtain the total scores for all 21 items. Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 is minimal depression, 14-19 is mild depression, 20-28 is moderate depression and 29-63 is severe depression.
Time Frame: Week 12 ± 2
Population: Validation analysis set of VADERA I population. Number of participants analyzed = participants with BDI-II score assessment at specified time-point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | VADERA I
Number analyzed (Participants) | 215
scores on a scale | 8.5 (7.8)
Statistical Analysis 1: Comparison: VADERA I; Number of participants analyzed (N) = 214; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Convergent Validity Criterion ρ > |0.50|; Spearman correlation coefficient = 0.71, 95% CI 2-sided [0.64 to 0.77] — Convergent correlation between BDI-II and MADRS

5. Primary Outcome: WHO-5 Index at Baseline: VADERA I
Description: WHO-5 questionnaire contains five items related to cheerfulness, calmness, feelings of vigor, feelings of being well rested after sleep, and personal interest. The respondent rated each question on a 6-point scale ranging from 0 ("at no time") to 5 ("all of the time") according to the proportion of time over the preceding 2 weeks that applied to the attribute in question. Scores were summated, with raw score ranging from 0 to 25. Then the scores were transformed to 0-100 by multiplying by 4, whereas 0 indicated the worst possible emotional well-being and 100 the best.
Time Frame: Baseline
Population: Validation analysis set of VADERA I population. Number of participants analyzed = participants with WHO-5 score assessment at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | VADERA I
Number analyzed (Participants) | 224
scores on a scale | 61.1 (23.6)
Statistical Analysis 1: Comparison: VADERA I; Number of participants analyzed (N) = 222; Test type: Superiority or Other; p = 0.034, t-test, 2 sided — Convergent Validity Criterion ρ > |0.50|; Spearman correlation coefficient = -0.59, 95% CI 2-sided [-0.67 to -0.49] — Convergent correlation between WHO-5 and MADRS
Statistical Analysis 2: Comparison: VADERA I; Number of participants analyzed (N) = 223; Test type: Superiority or Other; p = 0.010, t-test, 2 sided — Convergent Validity Criterion ρ > |0.50|; Spearman correlation coefficient = -0.61, 95% CI 2-sided [-0.68 to -0.52] — Convergent correlation between WHO-5 and BDI-II
Statistical Analysis 3: Comparison: VADERA I; Number of participants analyzed (N) = 222; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Convergent Validity Criterion ρ > |0.50|; Spearman correlation coefficient = -0.73, 95% CI 2-sided [-0.78 to -0.66] — Convergent correlation between WHO-5 and PHQ-9

6. Primary Outcome: WHO-5 Index at Week 12 ± 2: VADERA I
Description: as for outcome 5
Time Frame: Week 12 ± 2
Population: Validation analysis set of VADERA I population. Number of participants analyzed = participants with WHO-5 score assessment at specified time-point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | VADERA I
Number analyzed (Participants) | 206
scores on a scale | 63.9 (23.6)
Statistical Analysis 1: Comparison: VADERA I; Number of participants analyzed (N) = 202; Test type: Superiority or Other; p = 0.219, t-test, 2 sided — Convergent Validity Criterion ρ > |0.50|; Spearman correlation coefficient = -0.54, 95% CI 2-sided [-0.63 to -0.43] — Convergent correlation between WHO-5 and MADRS
Statistical Analysis 2: Comparison: VADERA I; Number of participants analyzed (N) = 199; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Convergent Validity Criterion ρ > |0.50|; Spearman correlation coefficient = -0.68, 95% CI 2-sided [-0.75 to -0.60] — Convergent correlation between WHO-5 and BDI-II
Statistical Analysis 3: Comparison: VADERA I; Number of participants analyzed (N) = 205; Test type: Superiority or Other; p < 0.001, t-test, 2 sided — Convergent Validity Criterion ρ > |0.50|; Spearman correlation coefficient = -0.77, 95% CI 2-sided [-0.82 to -0.70] — Convergent correlation between WHO-5 and PHQ-9

7. Primary Outcome: MADRS at Baseline: VADERA I
Description: The MADRS, an interview addressing 10 characteristics of depressive symptomatology, was used as the gold standard. The symptom-related information provided by each participant was rated on item-specific scales ranging from 0 (best) to 6 (worst) in order to evaluate individual symptom severity. Total score was sum of 10 characteristics, ranging from 0 to 60; 0, no depression; 60, severely depressed. Sum scores exceeding 12 indicated clinical relevance suggested mild to severe symptomatology.
Time Frame: Baseline
Population: Validation analysis set of VADERA I population. Number of participants analyzed = participants with MADRS assessment at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | VADERA I
Number analyzed (Participants) | 259
scores on a scale | 7.3 (6.4)

8. Primary Outcome: MADRS at Week 12 ± 2: VADERA I
Description: The MADRS, an interview addressing 10 characteristics of depressive symptomatology, was used as the gold standard. The symptom-related information provided by each participant was rated on item-specific scales ranging from 0 (best) to 6 (worst) in order to evaluate individual symptom severity. Total score was sum of 10 characteristics, ranging between 0 to 60; 0, no depression; 60, severely depressed. Sum scores exceeding 12 indicated clinical relevance suggested mild to severe symptomatology.
Time Frame: Week 12 ± 2
Population: Validation analysis set of VADERA I population. Number of participants analyzed = participants with MADRS assessment at specified time-point.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | VADERA I
Number analyzed (Participants) | 218
scores on a scale | 6.8 (6.3)

9. Primary Outcome: PHQ-9 Summary Score: VADERA II
Description: as for outcome 2
Time Frame: Baseline
Population: Full analysis set of VADERA II population defined as all study participants diagnosed with RA, who had given informed consent, and had completed at least one of the depression questionnaires. Number of participants analyzed = participants with PHQ-9 summary score assessment at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | VADERA II
Number analyzed (Participants) | 975
scores on a scale | 6.0 (4.7)

10. Primary Outcome: BDI-II Summary Score: VADERA II
Description: as for outcome 4
Time Frame: Baseline
Population: Full analysis set of VADERA II population. Number of participants analyzed = participants with BDI-II summary score assessment at baseline.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | VADERA II
Number analyzed (Participants) | 971
scores on a scale | 10.1 (8.8)

11. Primary Outcome: Percentage of Participants With Prevalence of Depressive Symptomatology Based on a BDI-II Score Greater Than or Equal to (≥)14 or PHQ-9 Score ≥5: VADERA II
Description: PHQ-9 is a self-reported questionnaire measuring depressive symptoms. This is a 9-item measure with a response score for each item on a 4-point scale ranging from 0 (not at all) to 3 (nearly every day). The total score ranges from 0 to 27; with 0-4 indicating no depressive symptoms, 5-9 mild, 10-14 moderate, 15-19 moderately severe, and 20-27 severe depression. BDI-II Scale is a 21-item self-reported questionnaire measuring existence and severity of depression symptoms. Symptoms are each scored on a 4-point scale of 0 (no symptom) to 3 (severe symptom). Total score ranges from 0-63; of which 0-8 is considered no depression, 0-13 minimal, 14-19 mild, 20-28 moderate, and 29-63 severe depression. Participants with a BDI-II score ≥14 or a PHQ-9 score ≥5 were classified as having depressive symptomatology. Participants were evaluated by positive depressive symptomatology for each questionnaire as well as being positive for both questionnaires combined or at least one of the questionnaires.
Time Frame: Baseline
Population: Full analysis set of VADERA II population.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | VADERA II
Number analyzed (Participants) | 1004
percentage of participants
  PHQ-9 score ≥5 | 55.1 [51.89 to 58.23]
  BDI-II score ≥14 | 27.7 [24.91 to 30.63]
  PHQ-9 score ≥5 or BDI-II score ≥14 | 55.4 [52.24 to 58.48]

ADVERSE EVENTS:
Time Frame: From Baseline to Week 12 ± 2
Arm/Group | VADERA I | VADERA II
Serious Adverse Events (participants affected / at risk) | 0/277 | 0/1015
Other Adverse Events (participants affected / at risk) | 0/277 | 0/1015

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.